CLINICAL TRIAL: NCT04946812
Title: Split-belt Treadmill Training to Rehabilitate Freezing of Gait and Balance in Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Alfonso Fasano, Clinician Investigator, Staff Neurologist, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-6049
Record Dates: First submitted 2021-06-12; First posted 2021-07-01 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease; Freezing of Gait; Gait, Unsteady
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Split-belt treadmill (Grail systems®, by Motek, Netherlands)
Who Masked: Outcomes Assessor
Masking Description: This is a prospective, single-blind, parallel-group randomized control trial to assess the feasibility and safety of SBTM in preventing falls and improving gait and balance, as well as its efficacy compared to TM training. The assessor will be blinded to their randomization. Patients will not be blinded to the intervention, and will be informed about the rationale of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The velocity of the belt will be adjusted to the over-ground speed of the subject, and will be reduced on the least affected side by 25%. While the speed of the treadmill will not change throughout the study, the duration of the training will increase each week. In the first week, the SBTM training will take place for 10 minutes. There will be a 5-minute rest period, and the split-belt conditions will continue for another 10 minutes of training (total training time= 20 minutes).
  Interventions: Other: Split-belt treadmill training
- Control group (Active Comparator): The subject will continue to walk under tied-belt conditions adjusted to the over-ground walking speed. In the first week, the treadmill training will be for 10 minutes. They will get a 5-minute break, similar to the intervention group, and continue for another 10 minutes under tied-belt conditions.
  The duration of each session will increase by 8 minutes every week. For example, in week 1, the treadmill training will be for a total of 20 minutes; in week 2, for 28 minutes; in week 3, for 36 minutes, and so forth, until it gets to 60 minutes by week 6. The rest period will remain at 5 minutes each session, and will always take place at the halfway mark. All 3 sessions in the week will have the same duration of training.
  If the subject cannot tolerate the velocity or duration of the session, the protocol will be adjusted to most recently tolerated session (and will be recorded for further interpretation and analysis).
  Interventions: Other: Split-belt treadmill training

INTERVENTIONS:
Other: Split-belt treadmill training — 18 sessions of SB-TM training, where the velocity of the belt will be adjusted to the over-ground speed of the subject, and will be reduced on the least affected side by 25%.

SUMMARY:
Parkinson's disease (PD) related gait and balance disorders are challenging to treat because they cannot be optimized with pharmacological intervention alone. This treatment gap is important to address because gait asymmetry and incoordination are associated with increased falls in this population, which can be functionally debilitating and lead to increased morbidity and mortality. Freezing of gait (FOG) has also been associated with reduced quality of life independent of its association with impaired mobility. Gait disorders therefore represent an unmet need in the treatment of PD. A split-belt treadmill (SB-TM) can be used to adjust the speed of each leg separately and individuals can be prompted to 'adapt' to an asymmetric gait and 're-adapt' with return to symmetrical gait in a phenomenon known as 'after-effect'.

DETAILED DESCRIPTION:
Parkinson's disease (PD) related gait and balance disorders are challenging to treat because they cannot be optimized with pharmacological intervention alone. This treatment gap is important to address because gait asymmetry and incoordination are associated with increased falls in this population, which can be functionally debilitating and lead to increased morbidity and mortality. Freezing of gait (FOG) has also been associated with reduced quality of life independent of its association with impaired mobility. Gait disorders therefore represent an unmet need in the treatment of PD.

Physiotherapy with treadmill training is a means to address the limitations of pharmacotherapy in this population. Treadmill training increases stride length, lowers cadence and improves foot clearance; long-term treadmill training results in clinically improved gait velocity and postural stability. The advent of SB-TM training can further optimize the gait instability that arises from asymmetric pathology in this population. The SB-TM has 2 belts, which can either move in unison (tied) or at different speeds (split), and it has been effective in restoring symmetrical gait in the stroke population, with gait adaptations retained for up to 3 months. The motor symptoms in PD develop asymmetrically, with the burden of symptoms often lateralizing to one side, so the SB-TM offers a unique opportunity to modulate spatial and temporal gait parameters to study gait adaptation in the PD population.

Split-belt treadmill training uses the concept of adaptive learning, which is error-driven motor leaning in response to changes in the external environment. It can be used to target specific gait deviations, and preliminary research has indicated that it can improve gait disorders in PD by decreasing limb asymmetry. Adaptive learning occurs when there is an adjustment of leg-speed perception during locomotor movement. When using a split-belt treadmill (SB-TM) to adjust the speed of each leg, the step length and double support time during gait can be manipulated. Individuals can therefore be prompted to 'adapt' to the asymmetric gait (e.g., the leg walking on a slow belt will take longer steps to accommodate to the leg walking on the faster belt) and 're-adapt' with return to symmetrical gait.

This method of rehabilitation can therefore be used to treat a range gait abnormalities and previous research has demonstrated the ability to restore symmetrical gait and reduced falls for up to 3 months in the stroke population. A preliminary study from our lab in individuals with PD and FOG demonstrated that velocity reduction by 25% on the least affected side resulted in a more symmetric and coordinated gait after 10 minutes of SB-TM training.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic PD
2. Hoehn & Yahr Stage 2-3, on levodopa
3. FOG, resistant to dopaminergic therapy
4. Disease duration: 5-15 years
5. Stable clinical response to medications or stimulation parameters (in case of DBS) for at least 3 months
6. MMSE >24/30
7. Able to walk on a motor-driven treadmill

Exclusion Criteria:

1. Severe imbalance that limits ambulation (Hoehn &Yahr score above 3)
2. Orthopedic conditions and other systemic disease affecting locomotion
3. Cardiac conditions limiting the ability to walk uninterrupted for 1 hour
4. Presence of other neurological disorder
5. Inability to be fluent in English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Falls | 3 months after completion of treadmill training
  The incidence of falls for 3 months after completing treadmill training. Falls will also be assessed at multiple stages during the 7.5-month study period, to understand the duration of benefit of this intervention. This data will be obtained from the falls calendar that will be provided to subjects upon their recruitment to the study.

SECONDARY OUTCOMES:
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Cadence (steps per minute)
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Stride time (time elapsed between the first contact of two consecutive footsteps of the same foot in milliseconds)
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Duration of stance (time during which the foot is in contact with the ground) o
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Swing (swing phase of gait begins when the foot first leaves the ground and ends when the same foot touches the ground again)
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Double limb support phase (he subperiod during which both feet are in contact with the ground)
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Step length, calculated by multiplying the 'step time' and 'belt speed'
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Step width height (the mediolateral space between the two feet)
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Kinemetics of joint excursion (expression as degree of range of motion)
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Foot angle (the angle made by the long axis of the foot from the heel to 2nd metatarsal and the line of progression of gait)
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Ratio of single support time/ double support time, which reflects dynamic stability
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Symmetry ratio (best leg step length/worst step)
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Coefficients of variation (which measures the variability of the temporal parameters of the swing phase duration and gait cycle time, and is represented by the (SD/mean) x100
Gait parameters between intervention and control groups | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Sequence effect (progressive reduction in step length), measured by a linear regression slope determined by plotting consecutive stride time intervals against stride number
Health-related quality of life | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Measured by the Parkinson's Disease Questionnaire-39 item self-report questionnaire (PDQ-39), scored out of 100 where a higher score reflects greater impact on quality of life
Balance and postural stability | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Measured by the Activities-specific Balance and Confidence (ABC) scale, possible range = 0 to 1600, Scores lower than 50 indicate a low level of functioning, scores above 50 but below 80 indicate a medium level, and those over 80 indicate a high level of functioning.
Freezing of gait | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Measured by the new freezing of gait questionnaire (NFOGQ).The total score ranges from 0 to 24, and higher scores denote more severe FOG.
Parkinson's disease signs and symptoms | Obtained at baseline evaluation, after 1.5 months of training, and 3-months post intervention
  Assessed by the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS). The maximum total UPDRS score is 199, indicating the worst possible disability from PD

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT04946812/Prot_000.pdf
  • Informed Consent Form (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT04946812/ICF_001.pdf